CLINICAL TRIAL: NCT05252039
Title: Goals in Focus: CBT for Motivational Negative Symptoms of Psychosis - a Randomized-controlled Feasibility Trial
Brief Title: Goals in Focus: CBT for Motivational Negative Symptoms of Psychosis
Acronym: GIF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Matthias Pillny, Trial Manager, University of Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRKS00018083
Record Dates: First submitted 2022-01-28; First posted 2022-02-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Psychosis; Schizophrenia; Negative Symptoms With Primary Psychotic Disorder
Keywords: Amotivation; Avolition; Anhedonia; Asociality
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Anhedonia

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, parallel-group, two-armed
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goals in Focus Therapy (Experimental): Participants in this arm will receive 24 weekly sessions with Goals in Focus therapy (GiF) over 6 months.
  Interventions: Behavioral: Goals in Focus
- Waitlist Control (No Intervention): Participants in this arm will not receive any psychological treatment for 6 months. After 6-months, they will receive 24 sessions of Goals in Focus Therapy.

INTERVENTIONS:
Behavioral: Goals in Focus — Goals in Focus (GiF) is a symptom-specific treatment program that targets motivational negative symptoms in patients with schizophrenia-spectrum disorders.
  The aim is to improve setting and pursuit of personal relevant goals.
  GiF follows a 24-individual-sessions treatment manual. GiF includes five treatment phases: 1) Preparation, 2) Goal-setting, 3) Goal-pursuit, and 4) Reflection and preparation of autonomous goal-pursuit. The interventions include generating positive goals, behavioral activation, training of anticipatory pleasure, challenging demotivating beliefs, training of problem-solving skills and social skills training.
  Arms: Goals in Focus Therapy

SUMMARY:
This pilot feasibility trial aims to evaluate the "Goals in Focus" intervention for motivational negative symptoms in people with psychosis.

Goals in Focus interventions translate findings of basic clinical research on psychological mechanisms of motivational negative symptoms into a tailored and comprehensive novel psychological treatment program.

The current single-blind randomized-controlled study aims to test feasibility and to examine first estimates of the expected effect size of Goals in Focus to inform a subsequent fully-powered RCT.

The feasibility data will be used to improve on the trial design and the provision of the "Goals in Focus" intervention where necessary.

DETAILED DESCRIPTION:
The reduction of goal-directed behavior is a core issue in motivational negative symptoms of psychosis and accounts for the long-term decline in psychological wellbeing and psychosocial functioning. However, the available treatment options are rather unspecific and show only small effects on motivational negative symptoms. Interventions that directly target the relevant psychological mechanisms of motivational negative symptoms are likely to be more effective. With "Goals in Focus", we translated findings of basic clinical research on psychological mechanisms of motivational negative symptoms into a tailored and comprehensive novel psychological treatment program for people with motivational negative symptoms. The current study aims to test the feasibility of Goals in Focus and trial procedures and 2) to estimate the expected effect size to inform a subsequent fully-powered trial.

A single-blind randomized-controlled trial will be conducted at the outpatient clinic of the Universität Hamburg, Germany. Thirty participants diagnosed with a psychotic spectrum disorder and at least moderate motivational negative symptoms will be randomly assigned to either 24 sessions of "Goals in Focus" or to a 6-months waitlist control group. Assessments will be conducted at baseline (t0) and 6 months after baseline completion (t1). Feasibility and acceptance of "Goals in Focus" will be rated by practitioners and participants. Feasibility of the trial procedures will be evaluated, e.g., with regard to patient recruitment, retention-, and attendance rates. The primary outcome for effect size estimation is defined as group differences in motivational negative symptoms at t1, corrected for baseline values. Secondary outcomes include psychosocial functioning, psychological well-being, depressive symptoms, expressive negative symptoms, negative symptom factors and goal-pursuit in everyday life.

The treatment effect on the primary outcomes will provide the basis for the sample size calculation for a fully powered RCT. The feasibility data will be used to improve on the trial design and the provision of the "Goals in Focus" intervention where necessary.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of a schizophrenia spectrum disorder (confirmed by the Structured Clinical Interview for DSM V Clinical Version
* at least moderate motivational negative symptoms (i.e., scores ≥ 3 (moderate) in two items or ≥ 4 (moderately severe) in one item of the 'motivation and pleasure factor' of the Brief Negative Symptom Scale (BNSS)
* sufficient skills in German language to participate in psychological therapy
* capable to engage in weekly therapy sessions of 50-minutes
* prioritize the reduction of negative symptoms as their current goal for treatment
* capable to give informed consent to participate in the trial

Exclusion Criteria:

* being at immediate and serious risk to self or others
* co-morbid diagnosis of alcohol or substance use disorder
* intake of Benzodiazepines for >2 days per week
* receiving any other psychological treatment aiming to reduce motivational negative symptoms

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Brief Negative Symptoms Scale (BNSS) - 'motivation and pleasure factor' score | 6 months after baseline assessment
  The primary outcome is defined as the change in motivational negative symptoms assessed with the 'motivation and pleasure factor' of the Brief Negative Symptoms Scale (BNSS). The BNSS is a 13-item semi-structured interview measuring negative symptoms on two factors, namely 'motivation and pleasure' and 'reduced expressivity'. The 'motivation and pleasure factor' includes seven items that measure the subscales of 'anhedonia', 'avolition', and 'asociality'. Symptoms are rated on a seven-point scale ranging from 0 "no impairment" to 6 "severe deficit"

SECONDARY OUTCOMES:
Avolition, Asociality and Anhedonia | 6 months after baseline assessment
  The respective subscales of the Brief Negative Symptom Scale according to the five-factor model. Each scale ranges from 0 to 6 with higher scores indicating higher symptom severity
Role Functioning Scale (RFS) | 6 months after baseline assessment
  Psychosocial Functioning across different domains of social roles
Global Assessment of Functioning (GAF) | 6 months after baseline assessment
  Observer-rating of psychosocial functioning. Ranges from 0 to 100 with higher scores indicating better functioning
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | 6 months after baseline assessment
  Self-reported psychological well-being. Scores range from 14 to 70 with higher scores indicating higher well-being
Calgary Depression Rating Scale for Schizophrenia (CDSS) | 6 months after baseline assessment
  Semi-structured interview ti assess depressive symptoms. Scores range from 0 to 36 with higher scores indicating more depressive symptoms
Goal-pursuit within daily-life | 6 months after baseline assessment
  Daily-life goal-pursuit will be assessed using the Experience Sampling Method (ESM). Participants will be prompted two times per day (10am and 10pm) over the course of one week via the MovisensXSapplication (Movisens GmbH) installed on a smartphone device. At the beginning of the ESM assessment, the participants' self-efficacy will be assessed with the Generalized Self-Efficacy Scale (GSE) Each of the following '10am prompts' will ask the participants to nominate a goal that they would like to achieve during the respective day and to rate characteristics of this goal (e.g., goal-commitment, goal-importance, goal-difficulty etc.). At the '10pm prompts', participants will be asked to indicate to what extent they achieved the respective goal and to answer questions on their causal-attributions and affective experience regarding their goal-achievement.

OTHER OUTCOMES:
Feasibility referrals | throughout the trial; approximately two years after recruitment commenced
  number of referrals (number of participants referred to the study)
Feasibility participant eligibility | throughout the trial; approximately two years after recruitment commenced
  eligibility rates (proportion of enrolled participants found eligible)
Feasibility consents | throughout the trial; approximately two years after recruitment commenced
  number of participants consenting to study participation and reasons for refusals
Feasibility retention | throughout the trial; approximately two years after recruitment commenced
  retention rate (i.e., number and proportion of participants who attend t1 assessment and completeness of data at t1)
Feasibility adherence | throughout the trial; approximately two years after recruitment commenced
  attendance rates and dose of intervention (i.e., number of sessions delivered within six months)
Feasibility data attrition | throughout the trial; approximately two years after recruitment commenced
  data attrition (proportion of outcome data not obtained)
Acceptability participants | throughout the trial; approximately two years after recruitment commenced
  - drop-out rate (i.e., number of withdrawals)
Acceptability and trial safety | throughout the trial; approximately two years after recruitment commenced
  - number of adverse and serious adverse events that are considered adverse reactions to the intervention
Treatment satisfaction participants | throughout the trial; approximately two years after recruitment commenced
  - participant satisfaction with treatment and personal outcomes (post-intervention questionnaire)
Treatment satisfaction therapists | throughout the trial; approximately two years after recruitment commenced
  - therapist satisfaction (post-intervention questionnaire therapist version)

CONTACTS AND LOCATIONS:
Overall Officials: Tania M Lincoln, Prof. Dr., Principal Investigator — Universität Hamburg
Locations (1):
- Psychotherapeutische Hoschschulambulanz Universität Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
only upon request

REFERENCES:
- [Derived] Schormann ALA, Pillny M, Hass K, Lincoln TM. "Goals in Focus"-a targeted CBT approach for motivational negative symptoms of psychosis: study protocol for a randomized-controlled feasibility trial. Pilot Feasibility Stud. 2023 May 2;9(1):72. doi: 10.1186/s40814-023-01284-4. PMID 37131247